CLINICAL TRIAL: NCT01071746
Title: The Predictive Utility of the Dimethylarginines and Ischemia Modified Albumin as Prognostic Biomarkers in Patients With Acute-on-chronic Liver Failure
Brief Title: Predictive Utility of DASIMAR as a Prognostic Biomarker in Acute-on-chronic Liver Failure (ACLF)
Acronym: DASIMAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Dr Rajeshwar P Mookerjee, University College London Hospitals
Other Study IDs: 08/HO714/8
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2010-02-19 (Estimated); Status verified 2008-04

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute decompensation of cirrhosis: acute decompensation of liver function occuring secondary to precipitating events such as sepsis, GI bleed.

SUMMARY:
Patients with acute on chronic liver failure have a risk of developing multiorgan failure and a high mortality. The current scoring systems defining the outcome of patients with acute decompensation of cirrhosis fail to identify patients that progress to Acute-on-chronic liver failure (ACLF).

The aim of the study is to evaluate if one can identify these patients early on with the proposed biomarkers: dimethylarginines and ischemia modified albumin.

DETAILED DESCRIPTION:
Patients with acute-on-chronic liver failure (ACLF) are at risk of multiorgan failure and high mortality. Recent data suggest that patients with decompensated liver cirrhosis have higher ADMA (asymmetrical dimethylarginine) levels compared to compensated cirrhosis and plasma ADMA levels correlate with severity of liver dysfunction and inflammation. There is also an increase in symmetric dimethylarginine (SDMA), a stereo-isomer of ADMA, which is largely excreted by the kidney. Plasma SDMA levels have been shown to be associated with patients

progressing to renal failure. In a pilot study by our group involving 52 patients with acute decompensation of chronic liver disease, we showed an increase in the summed product of ADMA and SDMA, which we termed dimethylarginine score ('DAS'): This was shown to have a good predictive utility for outcome in this small group of patients (AUROC=0.89).

Furthermore, we and others have shown that albumin of patients with advanced liver disease has widespread abnormalities. The amount of albumin that is found to have reduced metal binding capacity as a consequence of oxidative damage is termed Ischemia Modified Albumin (IMA).

Our data shows that patients with ACLF who die have a significantly increased IMA/serum albumin ratio (IMAR). The summation of these two pathologically relevant biomarkers (DAS+IMAR) we termed DASIMAR and found this score to have a better predictive utility than DAS alone (AUROC:0.91).

Primary objective : To identify the patients early on that progress to ACLF which would facilitate a goal directed therapeutic approach.

Secondary objective : Generation of this dataset will further define and enable prognostication of ACLF. If this study reveals a role for these biomarkers in patients with ACLF, commercial development of simple kits may be possible.

ELIGIBILITY:
Inclusion Criteria:

* All patients with an acute clinical decompensation of presumed cirrhosis (elevated bilirubin >85 µmol/L, or/and increasing ascites or/and hepatic encephalopathy < grade 2) related to a clear precipitating event (e.g. infection, bleeding, alcoholic hepatitis, exposure to hepatotoxin)

Exclusion Criteria:

* Admission for reasons other than decompensation of cirrhosis (other co-morbid diseases, especially established cardiovascular or renal disease (U/S).
* Malignancy (extra-hepatic or a hepatocellular carcinoma).
* Patients who have undergone major surgery or have unsolved surgical problems.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients with acute clinical deterioration of cirrhosis.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Progress to ACLF | hours, days

SECONDARY OUTCOMES:
Prognosticate ACLF | Days

CONTACTS AND LOCATIONS:
Overall Officials: Rajeshwar P Mookerjee, BScMRCPPhD, Principal Investigator — University College London Hospital
Locations (1):
- University College London Hospital, London, United Kingdom